CLINICAL TRIAL: NCT07275476
Title: Fibrin Clot Properties and Thrombin Generation in Pregnancy Women With and Without Obstetric Complications.
Brief Title: Pregnancy and Fibrin Clot Properties
Status: Recruiting | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Magdalena Piróg, MD, Principal Investigator, Jagiellonian University
Other Study IDs: 1072.6120.23.2025
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Fibrin Blood Clot; Pregnancy; Pregnancy Complicated by Cardiovascular Disorders as Postpartum Condition, Delivered During Previous Episode
Keywords: fibrinolysis; fibrin clot; thrombin generation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood samples will be drawn from an antecubital vein with minimal stasis using atraumatic venipuncture at 8 to 10 AM and collected into serum tubes and into tubes with anticoagulants: EDTAand sodium citrate (2.6 ml and 3.2%, respectively, 9:1) (Monovette, all from Sarstedt, Nümbrecht, Germany).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy pregnant women: Determination of fibrin clot properties and thrombin generation
  Interventions: Diagnostic Test: analysis of fibrin clot properties and thrombin generation
- Pregnant women with hypertensive disorders during pregnancy: Determination of fibrin clot properties and thrombin generation
  Interventions: Diagnostic Test: analysis of fibrin clot properties and thrombin generation

INTERVENTIONS:
Diagnostic Test: analysis of fibrin clot properties and thrombin generation — determination of fibrin clot properties and thrombin generation

SUMMARY:
1. The structure of fibrin clot and thrombin generation may vary between trimesters of pregnancy.
2. Unfavorably altered fibrin clot properties along with enhanced thrombin generation may lead to the development of complications during pregnancy such as TE and hypertensive disorders.
3. The application of machine learning techniques may help to identify previously undetected phenotypes with increased risk of TE and hypertensive disorders during pregnancy.

DETAILED DESCRIPTION:
Taken together, the integration of both fibrin clot properties and thrombin generation markers in pregnant women using modern science techniques may reveal new mechanisms explaining the relationship between altered fibrin clot properties and certain pregnancy complications. Moreover, it may help to identify new clot phenotypes of potential clinical significance, indicating prothrombotic risk or elevated chance of development of hypertensive disorders during pregnancy.

Specific working hypotheses:

1. The structure of fibrin clot and thrombin generation may vary between trimesters of pregnancy.
2. Unfavorably altered fibrin clot properties along with enhanced thrombin generation may lead to the development of complications during pregnancy such as TE and hypertensive disorders.
3. The application of machine learning techniques may help to identify previously undetected phenotypes with increased risk of TE and hypertensive disorders during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

I. age 18-40 years; II. natural conception (without assisted reproductive techniques).

Exclusion Criteria:

I. use of hormonal therapy (i.e., oral contraceptives, progestogens) within 3 months before or during pregnancy; II. use of anticoagulants oral/subcutaneous within 3 months before or during pregnancy; III. increased risk factors of VTE (i.e., obesity - body mass index >30 kg/m2; smoking) or history of VTE; IV. Concomitant diseases, i.e: severe hypertension, diabetes mellitus, autoimmune diseases (i.e., systemic lupus erythematosus, antiphospholipid syndrome); V. congenital or acquired thrombophilia (i.e., mutation factor V Leiden, prothrombin mutation).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females as they can get pregnant
Study Population: Two groups:
  1. Healthy pregnant women
  2. Pregnant women with hypertensive disorders during pregnancy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Fibrin clot phenotype | 12 months
  Fibrin clot phenotype

CONTACTS AND LOCATIONS:
Locations (1):
- Gynecological Endocrinology Department, Krakow, Małopolska, Poland

IPD SHARING:
Plan to Share IPD: No